CLINICAL TRIAL: NCT07220005
Title: Low Intensity Focused Ultrasound Stimulation in Stroke Patients - Parameter Optimization
Acronym: LIFUS-OPTIMIZE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00117400
Record Dates: First submitted 2025-10-21; First posted 2025-10-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Arm Weakness as a Consequence of Stroke; Upper Extremity Hemiparesis; Upper Extremity Impairments; Upper Extremity Weakness
Keywords: Brain Stimulation; Transcranial Focused Ultrasound Stimulation; Low Intensity Focused Ultrasound Stimulation; Stroke Recovery; Motor Learning; Corticospinal Excitability
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (6):
- ISPPA- 8 W/cm^2 (estimated intracranial spatial-peak pulse-average intensities) (Experimental): Participant will receive ultrasound stimulation at intensity of 8 W/cm^2 (estimated intracranial spatial-peak pulse-average intensities, ISPPA).
  Interventions: Device: Low intensity focused ultrasound stimulation
- ISPPA- 4 W/cm^2 (estimated intracranial spatial-peak pulse-average intensities) (Experimental): Participant will receive ultrasound stimulation at intensity of ISPPA of 4 W/cm^2
  Interventions: Device: Low intensity focused ultrasound stimulation
- Experimental: ISPPA- 0 W/cm^2 (estimated intracranial spatial-peak pulse-average intensities) (Sham Comparator): Participant will receive ultrasound stimulation at ISPPA- 0 W/cm^2 or sham stimulation
  Interventions: Device: Low intensity focused ultrasound stimulation
- Pulse repetition frequency(PRF) at 2000 Hz (Experimental): each participant will receive LIFUS with pulse repetition frequency at 2000 Hz
  Interventions: Device: Low intensity focused ultrasound stimulation
- Pulse repetition frequency(PRF) at 1000 Hz (Experimental): each participant will receive LIFUS with pulse repetition frequency at 1000 Hz
  Interventions: Device: Low intensity focused ultrasound stimulation
- Pulse repetition frequency (PRF) at 500 Hz (Experimental): Participants will receive LIFUS with pulse repetition frequency at 500 Hz
  Interventions: Device: Low intensity focused ultrasound stimulation

INTERVENTIONS:
Device: Low intensity focused ultrasound stimulation — A low-intensity focused ultrasound stimulation

SUMMARY:
The goal of this research study is to optimize the parameter of Low-Intensity Focused Ultrasound Stimulation (LIFUS) that is most effective in changing cortical excitability and motor learning skills in patients who suffered a stroke. The researchers hope to answer two questions.

* with increasing power, would LIFUS be more effective?
* with the same power, what LIFUS timing is the best

For Aim 1, the study will compare 8, 4 W/cm^2 to a zero(sham) stimulation to see if higher power is the better.

For Aim 2, the study will compare 500 vs 1000 vs 2000 Hz "timing" to see which one is better.

ELIGIBILITY:
Inclusion Criteria:

* age >=21 years old of any gender or race
* First-ever ischemic or hemorrhagic stroke (neuroimaging verified) at least 6 months from the stroke onset of symptoms
* Unilateral arm weakness measured by the Fugl-Meyer Upper-Extremity Scale ≤ 62/64
* Inducible rest motor threshold and testing motor threshold recorded from the affected abductor pollicis brevis muscle

Exclusion Criteria:

* Bilateral strokes (infarcts and/or hematoma)
* Other co-existent neuromuscular disorders affecting upper extremity motor impairment
* History of medically uncontrolled depression or other neuropsychiatric disorders despite medications either before or after a stroke that may affect the subject's ability to participate in the study
* History of confirmed dementia or taking dementia drugs
* Uncontrolled hypertension despite medical treatment(s) at the time of enrollment, defined as SBP≥185 mmHg or DBP≥110 mmHg (patient can be treated, reassessed and enrolled later)
* Presence of any MRI/TMS/LIFUS risk factors
* Concurrent enrollment in another interventional stroke recovery study
* Concerns that the subject cannot comply with study procedures and visits
* Pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Motor sequence learning | Baseline, immediately after intervention, and 1 hour after intervention
  Motor sequence learning (MSL) involves predictive processing that results in the anticipation of each component of a sequence of actions. MSL will produce response times and the MSL measure will be the number of responders (i.e., those with ≥20% reduction in the response time).
Corticospinal excitability | Baseline, immediately after intervention, and 1 hour after intervention.
  Corticospinal excitability is measured by the peak to peak amplitude of motor evoked potential.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Feng, MD MS, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No